CLINICAL TRIAL: NCT05361239
Title: Delayed Antibiotic Therapy in General Practice : Example of Acute Otitis Media in Adults and Children Over 6 Months of Age
Brief Title: Delayed Antibiotic Therapy in General Practice
Acronym: ADOMA
Status: Completed | Type: Observational
Sponsor: CNGE Conseil (Other)
Responsible Party: Sponsor
Other Study IDs: CNGE-2021/03; 2022-A00377-36 (Other: IDRCB)
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: AOM - Acute Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction In 2019, France was the 4th highest consumer of antibiotics in Europe. Among the interventions proposed to reduce antibiotic prescribing, delayed prescribing deserves particular attention. The effectiveness of delayed antibiotic prescription in reducing antibiotic consumption remains poorly studied in the literature, and no study has yet been conducted in France. The main objective of our study is to investigate the factors associated with the choice of antibiotic strategy(immediate or deferred). The secondary objectives are to study the frequency and factors associated with antibiotic consumption according to the initial prescription, and to determine the typical profiles of patients, in the context of a delayed prescription, who consume the antibiotic outside the GP's recommendations.

Method More 330 general practitioners in France will recruit 2800 patients older than 6 months with acute otitis media between September 2022 and April 2023. GPs will be recruited via the CNGE investigator network, the colleges of general medicine in Ile-de-France, the Sentinelles network, the French Medical Association and the regional unions of health professionals.

Initial medical data will be collected by the physicians. Patients will fill in daily data for 2 weeks to monitor their disease. They will also fill in social data, and questionnaires assessing their level of health literacy, confidence and satisfaction with the general practitioner consulted.

Factors associated with the physician's choice of antibiotic therapy and the patients' consumption of antibiotics will be analyzed via mixed models. Consumption rates will be expressed as percentages with their confidence intervals.

Conclusion This work will allow a better understanding of the elements that guide physicians towards delayed prescription. It can help physicians to better assess patients who are likely to be non-compliant with delayed prescription in order to avoid this type of prescription for them.

DETAILED DESCRIPTION:
In 2018, France was the third country in Europe for antibiotic consumption. Each year, 33,000 deaths in Europe, from which 12,500 in France, could be due to antibiotic-resistant bacteria . Without changes in practice, antibiotic-resistant bacteria could be responsible for more than 10 million deaths worldwide by 2050.

In France, Général Practitioners (GP) are responsible for most antibiotic prescriptions and 2nd prescribers in Europe. The annual cost of antibiotic overconsumption, in primary care, is estimated between 71 and 442 millions euros. Otolaryngology's infections are responsible for 44% of these prescriptions. While antibiotic consumption has been declining since 2000, the situation seems to be reversing since 2010 with an increase of 5.6% between 2011 and 2016.

Several interventions on GP's have been evaluated to reduce antibiotic use, but none seemed to prove a mid/long term efficacy. Patient interventions combined with physician interventions appear to be more effective. Delayed antibiotic prescribing (DAP), a method of delaying the filling of an antibiotic prescription for at least 48 hours, deserves special attention. The effectiveness of DAP in reducing antibiotic consumption remains poorly studied in the literature, and no study has yet been conducted in France. Physicians consider acute otitis media to be the most appropriate condition for PDA, mainly because of doubts about the value of antibiotics in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 6 months
* At least one of the following signs:

  * moderate to severe tympanic membrane bulge or recent onset of otorrhea not caused by otitis externa,
  * mild tympanic membrane bulge associated with either:

    * recent onset (less than 48 hours) of otalgia (or holding, pulling, rubbing the ear in a child who does not speak) or,
    * tympanic erythema
* Enrolled in a social security plan or beneficiary of such a plan.
* Patient who has given oral non-objection after being fully informed about the protocol.

Exclusion Criteria:

* - AOM in the previous 3 months or recurrent AOM (≥ 3 in 6 months or ≥ 4 in 12 months)
* Presence of paracentesis tubes or perforated tympanic membrane
* Acute complication of otitis (mastoiditis, meningitis, intracranial abscess, sinusal thrombosis or facial nerve paralysis)
* Additional intercurrent bacterial infection such as diagnosed or suspected pneumonia
* Symptomatology that suggests a more serious condition to the clinician
* Hospitalization or emergency care required
* Patients at risks of complication (immunosuppression)
* Associated severe acute pathology
* Cranio-facial malformation, down syndrom, cystic fibrosis
* Antibiotic therapy in the previous seven days
* Minor patient not accompanied by a legal representative (father or mother)
* Patients already included in the study
* Patients who does not speak french
* Person subject to a legal protection measure
* Persons deprived of liberty
* Pregnant women, parturients and breastfeeding mothers

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Minors and adults consulting a GP for AOM
Sampling Method: Non-Probability Sample
Enrollment: 865 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
To study associated factors (GPs, patients, severity of illness) with the choice of antibiotic strategy (immediate or delayed, when antibiotic was prescribed). | At 14 days after inclusion
  Identification of associated factors (GPs, patients, severity of illness) with the choice of antibiotic strategy (intial or delayed) when antibiotic was prescribed

SECONDARY OUTCOMES:
Study the factors associated with no antibiotic prescription | At 14 days after inclusion
  Identification of associated factors with no antibiotic prescription
Describe the frequency of each strategy in our study sample | At 14 days after inclusion
  Frequencies of each antibiotic strategy used by GPs (initial antibiotic, delayed antibiotic, no antibiotic) in our sample of GPs
Describe the frequency of antibiotic use by patients according to choice of antibiotic strategy. | At 14 days after inclusion
  Frequencies of antibiotic consumption by patients according to the choice of antibiotic strategy (immediate, delayed or absent)
Describe factors associated with antibiotic consumption | At 14 days after inclusion
  Frequencies of antibiotic consumption by patients.
  In case of delayed antibiotic prescription, frequencies of antibiotic consumption by patients :
  * According to GP's recommandation
  * In spite of GP's recommandation
Determine a typical profile of patients using antibiotics outside of their GP's recommendations in case of delayed antibiotic prescription | At 14 days after inclusion
  Identification of the different patient factors associated with antibiotic consumption, and more specifically with the use of antibiotics in spite of GP's recommendations, in order to define a typical profile

CONTACTS AND LOCATIONS:
Locations (1):
- MSPU Jacques Prévert10 place George Sand, Montigny-le-Bretonneux, France